CLINICAL TRIAL: NCT05806840
Title: Enhancing the Impact of Evidence-Based Prevention for Youth: The Rapid Adaptation to Prevent Drug Use (RAPD) Implementation Study
Brief Title: Rapid Adaptation to Prevent Drug Use
Acronym: RAPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andria B Eisman, Assistant Professor of Community Health, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-23-01-5434; R34DA056777 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-04-10 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Michigan Model for Health (MMH) Curriculum Implementation (Active Comparator): Standard implementation of the MMH (Michigan Model for Health), a universal prevention intervention includes curriculum materials, foundational curriculum training and as-needed technical assistance, provided by the regional school health coordinators.
  Interventions: Behavioral: Standard Implementation
- Rapid Adaptation to Prevent Drug Use (RAPD) (Experimental): RAPD is a novel bundle of implementation strategies to improve the responsiveness of an existing evidence-based intervention (EBI), the Michigan Model for Health (MMH) for urgent drug events. These implementation strategies will be deployed in addition to standard implementation components.
  Interventions: Behavioral: Rapid Adaptation to Prevent Drug Use (RAPD)

INTERVENTIONS:
Behavioral: Rapid Adaptation to Prevent Drug Use (RAPD) — RAPD will include a novel bundle of implementation strategies to support rapid responses to urgent drug use events. The strategies deployed will be based on the first step of the After Action Review: critical analysis and reflection.
  Arms: Rapid Adaptation to Prevent Drug Use (RAPD)
Behavioral: Standard Implementation — Standard implementation of the Michigan Model for Health (MMH) includes curriculum materials and as-needed technical assistance provided by a school health coordinator.
  Arms: Standard Michigan Model for Health (MMH) Curriculum Implementation

SUMMARY:
Using a 2-group, mixed method cluster randomized trial design, this study will compare standard implementation versus RAPD implementation strategy in Michigan Middle Schools

DETAILED DESCRIPTION:
Background: Drug use trends change rapidly among youth, leaving intervention experts struggling to respond to emerging drugs promptly. There is a critical need to advance implementation strategies to optimize system responsiveness to these emerging issues. COVID-19 has increased the urgency for implementation science to facilitate rapid, equitable responses using existing treatment and prevention efforts. Tier 1 evidence-based interventions (EBIs), such as the Michigan Model for Health™ (MMH) lend themselves to addressing emerging trends. The overall objectives of this study are to 1) improve the responsiveness of school-based EBIs in addressing urgent issues and 2) find ways to support educators and education systems in implementing updated EBIs, attending to unique considerations of low-resource settings.

Methods: Using a 2-group, mixed method, randomized controlled trial design, this pilot study will compare standard implementation versus the RAPD implementation strategy to deliver MMH.

The RAPD implementation strategy was designed based on an After Action Review (AAR) approach in collaboration with community partners to analyze gaps and best practices and identify and test suitable implementation strategies to improve responsiveness to the next urgent drug event.

ELIGIBILITY:
Inclusion Criteria:

* Schools that fail to meet state standards for implementation (less than 80% of curriculum) and/or face one or more barriers to Michigan Model for Health (MMH) curriculum implementation
* Schools that have a minimum of 25% of students eligible for free and reduced meals
* Schools must include 7th-grade classes/students

Exclusion Criteria:

* Schools that meet state identified fidelity standards (i.e., teaching 80% or more of the curriculum) and do not face barriers to MMH implementation
* Schools that have fewer than 25% of students eligible for free and reduced meals
* Schools that do not include 7th-grade education level

Ages: 11 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
RAPD Strategy Feasibility | 9 Months
  The investigators use a mixed methods approach to determine teacher perceived feasibility of the RAPD implementation strategy (Feasibility of Implementation Measure). Feasibility is defined as the extent to which the innovation (RAPD) can be practically used in a given setting.
RAPD Strategy Acceptability | 9 Months
  The investigators use a mixed methods approach to determine teacher perceived acceptability of the RAPD implementation strategy (Acceptability of Implementation Measure). Acceptability is defined as the view among stakeholders that a given innovation (RAPD) is agreeable or satisfactory.
RAPD Strategy Appropriateness | 9 Months
  The investigators use a mixed methods approach to determine teacher perceived appropriateness of the RAPD implementation strategy (Implementation Appropriateness Measure). Appropriateness is defined as the perceived compatibility of an innovation (RAPD) with needs and practices of the setting and the perceived utility in addressing a given problem.

SECONDARY OUTCOMES:
MMH Fidelity | 9 Months
  The investigators use an MMH fidelity tracking form to assess dose delivered by summing the total lessons delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Andria Eisman, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Wiltsey Stirman S, Baumann AA, Miller CJ. The FRAME: an expanded framework for reporting adaptations and modifications to evidence-based interventions. Implement Sci. 2019 Jun 6;14(1):58. doi: 10.1186/s13012-019-0898-y. PMID 31171014
- [Derived] Eisman AB, Koffkey C, Brown S, Holmes C, Schmidt B, Swihart E, Robinson T, Kim B. Using After Action Review to Identify Rapid Response Implementation Strategies for Emerging Drugs Among Youth. Prev Sci. 2025 Feb;26(2):258-270. doi: 10.1007/s11121-025-01787-x. Epub 2025 Feb 10. PMID 39930106
- [Derived] Eisman AB, Koffkey C, Partridge RT, Brown S, Kim B. Rapid Adaptation to Prevent Drug Use (RAPD): protocol of a pilot randomized trial to enhance the impact of an evidence-based intervention for youth. Pilot Feasibility Stud. 2025 Jan 21;11(1):8. doi: 10.1186/s40814-024-01581-6. PMID 39838453